CLINICAL TRIAL: NCT06497816
Title: An Investigation of Health Literacy, Physical and Cognitive Function, Health-related Behaviors, and Quality of Life in Chronic Obstructive Pulmonary Disease and Healthy Individuals
Brief Title: Health Literacy, Physical and Cognitive Function, Health-related Behaviors, and Quality of Life in COPD
Status: Recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Aslihan Cakmak, Principal Investigator, Hacettepe University
Other Study IDs: SBA24/414
Record Dates: First submitted 2024-06-28; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: COPD; Health Literacy; Health-Related Behavior
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Health Behavior

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COPD: Individuals with stable COPD
  Interventions: Other: No intervention
- Healthy Individuals: Healthy controls
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Health literacy is important for controlling disease progression and living a healthy life with illness. High health literacy is associated with higher cognitive performance and lower health-related quality of life. Physical, psychological, and social impairments are seen in chronic obstructive pulmonary disease (COPD). Studies investigating the relationship between health literacy and functional capacity, quality of life, physical activity, cognitive function, health-related behavior, and activities of daily living in individuals with COPD are limited. Therefore, the aim of this study was to compare individuals with COPD with healthy individuals in terms of health literacy, functional capacity, quality of life, physical activity, cognitive function, health-related behavior, and activities of daily living and to investigate the relationship between health literacy and functional capacity, quality of life, physical activity, cognitive function, health-related behavior, and activities of daily living in individuals with COPD.

ELIGIBILITY:
Inclusion criteria for the COPD group:

* Being over 40 years old,
* Diagnosed with COPD and being clinically stable,
* Being able to cooperate with the tests to be performed,
* Not having any cardiovascular disease, orthopedic or neurological problems that may affect the tests,
* Being willing to participate in the study.

Exclusion criteria for the COPD group:

* Being in an acute exacerbation period,
* Having any cardiovascular disease, orthopedic or neurological problems that may affect the tests,
* Not being willing to participate in the study.

Inclusion criteria for the control group:

* Being willing to participate in the study and being over 40 years old
* Not having any known disease

Exclusion criteria for the control group:

* Not being able to cooperate with the tests to be performed
* Not being willing to participate in the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with COPD and Healthy Controls
Sampling Method: Probability Sample
Enrollment: 144 (Estimated)
Dates: Start 2024-06-15 (Actual); Primary Completion 2027-06-15 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Functional capacity | 1st day
  Functional capacity assessment using self-paced 6-minute walk test.
Health literacy | 1st day
  Test of Functional Health Literacy in Adults will be used to evaluate health literacy. The TOFHLA is scored on a scale of 0 to 100 and higher scores indicate higher health literacy.
Health literacy | 1st day
  The Rapid Estimate of Adult Literacy in Medicine questionnaires will be performed. A score of 59 or less is defined as indicating low health literacy and a score of 60 or more indicates adequate health literacy.
Cognitive function | 1st day
  Montreal Cognitive Assessment will be used to evaluate cognitive function. The Montreal Cognitive Assessment scores range between 0 and 30. A score of 26 or over is considered to be normal.
Health-related behavior | 1st day
  Health-related Behavior Scale II will be performed to assess health-related behavior. The Health-related Behavior Scale II measures various health-related behaviors and is designed to assess the frequency or extent of engagement in these behaviors. Higher scores of the scale indicate more frequent or healthier behaviors, depending on the specific behavior being measured.
Functional exercise capacity | 1st day
  One-minute sit to stand test will be performed. The number of repetitions will be recorded.

SECONDARY OUTCOMES:
Forced vital capacity | 1st day
  Pulmonary function test using a spirometer will be performed. Forced vital capacity will be recorded.
Forced expiratory volume in one second | 1st day
  Pulmonary function test using a spirometer will be performed. Forced expiratory volume in one second will be recorded.
forced expiratory volume in one second/forced vital capacity ratio | 1st day
  Pulmonary function test using a spirometer will be performed. Forced expiratory volume in one second/forced vital capacity ratio will be recorded.
Peak expiratory flow | 1st day
  Pulmonary function test using a spirometer will be performed. Peak expiratory flow will be recorded.
Forced mid-expiratory flow (FEF25-75) | 1st day
  Pulmonary function test using a spirometer will be performed. Forced mid-expiratory flow (FEF25-75) will be recorded.
Physical activity level | 1st day
  Physical activity will be evaluated with International Physical Activity Questionnaire questionnaire. The questionnaire assesses physical activity across different domains, including leisure time, domestic and gardening activities, work-related activities, and transport-related activities. Scores are calculated based on the duration (minutes) and frequency (days) of these activities over the past seven days. Higher scores on the IPAQ indicate a higher level of physical activity.
Assessment of quality of life | 1st day
  St. George quality of life questionnaire will be used to assess quality of life. Higher scores reflect worse health status.
Activities of daily living | 1st day
  Activities of daily living will be evaluated using Leicester Cough Questionnaire. Each question is scored on a scale from 1 (maximum impact) to 7 (minimal impact). An average score is calculated for each domain (physical, psychological, and social), resulting in scores ranging from 1 to 7 per domain, and a total score between 3 and 21. A higher score indicates less impact.
Assessment of quality of life | 1st day
  Short Form-36 will be applied for assessing quality of life. Higher scores indicate better health status.

CONTACTS AND LOCATIONS:
Overall Officials: Aslihan Cakmak-Onal, PhD, PT, Principal Investigator — Hacettepe University; Deniz Inal-Ince, PhD, PT, Study Director — Hacettepe University; Elif Kocaaga, MSc, PT, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University Faculty of Physical Therapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No